CLINICAL TRIAL: NCT02580903
Title: Pulmonary Hypertension in Patients With Philadelphia Chromosome Negative Myeloproliferative Neoplasms; an Observational Prospective Study
Brief Title: Pulmonary Hypertension in Patients With Myeloproliferative Neoplasms
Acronym: MPNPH
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mette Brabrand, Staff Specialist, Odense University Hospital
Other Study IDs: MPNPH
Record Dates: First submitted 2015-01-31; First posted 2015-10-20 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Myeloproliferative Disorders; Pulmonary Hypertension
MeSH Terms: conditions — Myeloproliferative Disorders; Hypertension, Pulmonary | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All patients will submit a blood sample for later analysis
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radiology — Only a small subsample will require CT and right heart catherisation

SUMMARY:
This is an observational prospective study aiming to clarify the prevalence of pulmonary hypertension in patients with Myeloproliferative Neoplasms and their prognosis.

All patients attending our department with the above mentioned neoplasms will be offered inclusion in this study. All will have an echo performed and patients identified as being at risk of pulmonary hypertension will be offered complete investigation as specified by the European Cardiology Association.

All patients will be followed up for a total of five years to identify prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Myeloproliferative Neoplasms (PV, ET, PMF according to WHO classification)

Exclusion Criteria:

* Pregnancy
* Lack of informed consent
* Age < 18 years
* Cognitive dysfunctions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending our outpatient clinic with Myeloproliferative Neoplasms
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-02; Primary Completion 2018-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of pulmonary hypertension at initial presentation and first echo | Initial recruitment

SECONDARY OUTCOMES:
Mortality | 1 and 5 years
Incidence of pulmonary hypertension while under follow-up | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mette Brabrand, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark